CLINICAL TRIAL: NCT06774976
Title: Efficacy and Acceptability of an Evidence-Based Neck Resistance Training Program on Head Acceleration and Isometric Neck Strength in Female Soccer Players: A Pilot Quasi-Experimental Trial
Brief Title: Effect of Neck Training on Outcomes Related to Sport-Related Concussion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MLP1033
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Sport-related Concussion
Keywords: Sport-related concussion; Neck muscles; Primary prevention; Resistance training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Resistance Training (Experimental): 8-week Evidence-Based Neck Resistance Training Program
  Interventions: Other: 8-week Evidence-Based Neck Resistance Training Program
- Training as Usual (No Intervention): Usual Training Regiment

INTERVENTIONS:
Other: 8-week Evidence-Based Neck Resistance Training Program — See arm/group description.
  Arms: Neck Resistance Training

SUMMARY:
Sport-related concussion (SRC) is a significant concern in soccer. This pilot quasi-experimental trial aims to investigate the efficacy and acceptability of an evidence-based neck resistance exercise program in female soccer athletes for SRC prevention. The 8-week intervention includes dynamic and static neck exercises designed to reduce linear and rotational head accelerations, improve neck muscle strength, and minimise SRC risk. The study will evaluate program outcomes through laboratory testing, questionnaires, and user feedback. Findings from this pilot study will inform the design and implementation of a full-scale study, aiming to advance preventive strategies in SRC and address the underrepresentation of female athletes in research.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and acceptability of a novel evidence-based neck resistance training program for female soccer players. The primary objective is to assess the program's impact on neck strength and head accelerations during impact, with the broader goal of informing strategies to reduce the risk of sport-related concussions in soccer. A pilot quasi-experimental design will be employed to test the intervention and collect preliminary data for future large-scale trials.

Two senior-level female soccer teams will be invited to participate in the study. One team will be allocated to the intervention group, while the other will serve as the control group. The intervention group will undertake an eight-week neck resistance training program designed according to current resistance training prescription guidelines. The program consists of both static and dynamic exercises implemented with a head harness and resistance tubing to allow variable resistance loads. To ensure flexibility and adherence, the program is designed to be conducted either during the team's regular on-field soccer training or off-field gym sessions. Participants will complete the exercises two to three times per week. The control group will continue their usual training practices without incorporating any neck-specific resistance training during the study period.

Before the intervention, participants from both teams will undergo comprehensive baseline testing at Lund University's Movement and Reality Lab (MoRe-Lab). The testing will include three main components: isometric neck strength testing, head acceleration testing, and muscle activation analysis. Neck strength will be assessed in four cervical directions-flexion, extension, lateral flexion, and rotation-using a handheld dynamometer. Athletes will be seated in a high-backed chair and secured with straps to isolate head and neck movement. A snugly fitted head harness will be connected to the dynamometer, and participants will be instructed to exert maximal force during three-second isometric contractions in each direction. Each athlete will perform three repetitions, and the highest force value recorded in newtons will be used for data analysis.

Head acceleration will be assessed using a custom-built device designed to measure safe, controlled head movements. Athletes will be seated in the device and strapped securely to ensure only head and neck movement is permitted. A head harness connected to a drop mechanism will deliver a one-kilogram weight drop from a height proportional to the athlete's stature. This will produce safe, measurable linear and rotational head accelerations, with head movement captured by the Qualisys motion capture system. Data from this system will be used to calculate both linear and rotational accelerations in all four cervical directions.

To evaluate muscle activation patterns during head acceleration testing, surface electromyography (EMG) sensors will be placed on the sternocleidomastoid muscles and the trapezius (pars descendens). These exploratory outcomes will provide additional insights into the neuromuscular responses elicited by the intervention.

Following the baseline assessments, teams will proceed to the intervention phase. After the eight-week intervention, participants will return for follow-up testing, which will replicate the baseline assessments. At the conclusion of the study, all players and coaches will complete a questionnaire designed to evaluate the acceptability of the exercise program. This questionnaire will include both Likert-scale items and open-ended questions, allowing participants to provide detailed feedback and suggest potential improvements to the program.

Data analysis will focus on comparing changes in key outcomes within and between the intervention and control groups. The primary outcomes-changes in isometric neck strength and head accelerations-will be analyzed using repeated measures analysis of variance (ANOVA). Secondary outcomes, including the acceptability data, will be analyzed descriptively for Likert-scale responses, while qualitative feedback from open-ended questions will undergo thematic analysis. Exploratory outcomes, such as muscle activation data, will be evaluated descriptively to assess activation patterns during head accelerations.

To ensure adequate statistical power, an a priori sample size calculation using G*Power (v. 3.1.9.7, Düsseldorf, Germany) determined that a minimum of 34 participants would be required for repeated measures ANOVA (effect size f > 0.25, power 0.80, α = 0.05). Adjusting for cluster randomization using a variance inflation factor with a moderate intracluster correlation coefficient (ρ = 0.05) and accounting for a 25% dropout rate, the target sample size increased to 96 participants. For this pilot study, approximately half of the required sample size-around 50 participants-will be enrolled across the two soccer teams. This approach ensures the safety and feasibility of the intervention, provides preliminary effect sizes, and informs the design of a future full-scale trial.

The research team includes Branimir Ivanic, PT, MSc, Anna Cronström, PT, PhD, Nicholas Ryan, PhD, and Professor Eva Ageberg, PT, PhD, all affiliated with Lund University, Sweden. Professor Ageberg serves as the Principal Investigator for the study.

ELIGIBILITY:
Inclusion Criteria:

* Teams that are located in Skåne county
* Teams that are trained by professional trainers who are financially compensated for their work
* Teams that are not engaged in any targeted neck-strengthening exercises during the trial period beyond those prescribed within the trial
* Players that are 16 years of age or older
* Players that regularly attend all senior-level team activities, including training and match sessions
* Players that free of any injuries to their upper or lower limbs, torso, neck, or head at the time of enrolment
* Players with no history of undiagnosed neck pain within the previous three months.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Linear head acceleration | Measurements will be taken at baseline and after the 8-week intervention program.
  Linear head accelerations will be assessed during impulsive loads applied to the head in four cervical directions: flexion, extension, lateral flexion, and rotation. The impulsive load will be induced using a custom-made device, and linear accelerations will be measured with a Qualisys motion capture system, reported in units of gravitational force (g-force).
Rotational head acceleration | Measurements will be taken at baseline and after the 8-week intervention program.
  Rotational head accelerations will be assessed during impulsive loads applied to the head in four cervical directions: flexion, extension, lateral flexion, and rotation. The impulsive load will be induced using a custom-made device, and rotational accelerations will be measured with a Qualisys motion capture system, reported in radians per second squared (rad/s²).
Isometric neck strength | Measurements will be taken at baseline and after the 8-week intervention program.
  Isometric neck strength measured in all four cervical directions (flexion, extension, lateral flexion, and rotation) using a handheld dynamometer and will be reported in Newtons (N).

SECONDARY OUTCOMES:
Acceptability of an evidence-based neck resistance training program | The questionnaire will be distributed to athletes and trainers at the end of the 8-week
  The questionnaire, which has been developed in accordance with the Theoretical Framework of Acceptability, consists of seven statements that athletes will rate on a 5-point Likert scale (1=strongly disagree; 5=strongly agree), as well as two open-ended questions.

OTHER OUTCOMES:
Neck Muscle Activation Timing | Measurements will be taken at baseline and after the 8-week intervention program.
  Surface EMG sensors will be positioned on the neck musculature to measure neck activation patterns during head acceleration tests. The sensors will capture the time of muscle onset relative to the onset of force application to the head, measured in milliseconds (ms).
Neck Muscle Activation Amplitude | Measurements will be taken at baseline and after the 8-week intervention program.
  Surface EMG sensors will be positioned on the neck musculature to measure neck activation patterns during head acceleration tests. The sensors will capture the amplitude of muscle activation, which will be reported as a percentage of the amplitudes measured during maximal voluntary isometric neck strength.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Lund University
Locations (1):
- MoRe Lab, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD for primary and secondary outcomes will be made available upon reasonable request.